CLINICAL TRIAL: NCT04970329
Title: Corneal Thickness Changes in Patient Undergoing Dry Eye Managment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Fatima Hussain, principal investigator, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUF/MPO/2102
Record Dates: First submitted 2021-06-10; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — polyethylene glycol 400

STUDY DESIGN:
Intervention Model Description: 96 eyes will be divided into 3 groups (32 eyes each) and will be provided intervention which is Polyethylene Glycol 400 0.4%-Propylene Glycol 0.3%. , Dextran 0.1%Hypromellose 0.3%, and placebo(normal saline)
Who Masked: Participant, Investigator
Masking Description: Both participant and investigator will be masked about the treatment options.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Systane (Experimental): Instill one drop three times a day for one month.
  Interventions: Drug: Polyethylene Glycol 400 0.4%-Propylene Glycol 0.3%. and Dextran 0.1%Hypromellose 0.3%,
- Tears Naturale 2 (Experimental): Instill one drop three times a day for one month.
  Interventions: Drug: Polyethylene Glycol 400 0.4%-Propylene Glycol 0.3%. and Dextran 0.1%Hypromellose 0.3%,
- Placebo (Placebo Comparator): Instill one drop three times a day for one month.
  Interventions: Drug: Polyethylene Glycol 400 0.4%-Propylene Glycol 0.3%. and Dextran 0.1%Hypromellose 0.3%,

INTERVENTIONS:
Drug: Polyethylene Glycol 400 0.4%-Propylene Glycol 0.3%. and Dextran 0.1%Hypromellose 0.3%, — Drugs will be given to two group and third group will kept on placebo.
  Other Names: Systane and Tears Naturale 2

SUMMARY:
The purpose of this research is to the determine effect of dry eye and to compare the effect of artificial tears on central and peripheral corneal thickness.

DETAILED DESCRIPTION:
In this randomized controlled trial, 96 eyes of females with dry eye will be recruited through random sampling. Dry eye assessments will be done including TBUT, Schirmer test 1, and OSDI questionnaire. 96 eyes will be divided into 3 groups (32 eyes each) and will be provided intervention which is Polyethylene Glycol 400 0.4%-Propylene Glycol 0.3%. , Dextran 0.1%Hypromellose 0.3%, and placebo(normal saline) through randomization by an unmasked investigator. Changes in central and peripheral corneal thickness will be evaluated by corneal topography. Patients will be evaluated at baseline, after 15 days, after 1 month, and re-evaluated after 1 month of cessation of treatment.

ELIGIBILITY:
Inclusion Criteria:

● Females with ages ranging between 18-40 years and OSDI scores greater than 13, ametropia of up to 1DS of SE with astigmatism of less than 0.5DC, and Emmetropes.

Exclusion Criteria:

* Refractive error of more than ±1 Ds of SE and astigmatism of greater than ±0.5DC.
* Corneal surface disease other than dry eye disease.
* Corneal ectasia.
* Corneal or eyelid infections
* Age < 18 and >40 years.
* History of contact lens wears within the past three months.
* Male will be excluded because sex has a large influence on the symptomatology of DED Males have significantly low symptom scores as compared to females.
* Corneal surgeries.
* History of ocular /systemic disease within the past 6 months.
* The patients already receiving any kind of treatment for DED and other ocular diseases.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Dry eye has more prevalence in females.
Enrollment: 96 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in Corneal Thickness in microns | one month
  effect of dry eye treatment on the thickness of the cornea in microns measured by using corneal topography.
Change in Corneal Thickness in microns after treatment discontinuation. | one month
  after on month of treatment discontinuation access the change in corneal thickness in microns by using corneal topography.

SECONDARY OUTCOMES:
Improvement in dry eye | one month
  after treatment with artifical tears improvement in the tear break-up time in seconds and schirmer test values in millimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Faisalabad, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No